CLINICAL TRIAL: NCT00867503
Title: Open Label Phase II Trial of Bendamustine Hydrochloride (HCL) in Women With Advanced Ovarian Cancer
Brief Title: Open Trial of Bendamustine Hydrochloride in Women With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1137-04
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; bendamustine
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bendamustine (Experimental): bendamustine HCL 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
  Interventions: Drug: Bendamustine HCL

INTERVENTIONS:
Drug: Bendamustine HCL — bendamustine HCL 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
  Other Names: bendamustine hydrochloride

SUMMARY:
The study design is a non-randomized, open label, single center Phase II trial. Eligible patients are women who have a confirmed diagnosis of ovary, fallopian tube cancer or primary peritoneal serous papillary carcinoma who have relapsed or are refractory to therapy after primary treatment of their disease.

Patients will be treated with bendamustine Hydrochloride 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2. 20 patients will be enrolled in the study.

OBJECTIVES Hypothesis/Rationale: To determine the efficacy and safety of bendamustine hydrochloride, in women with platinum and taxane refractory ovarian cancer.

DETAILED DESCRIPTION:
Bendamustine, a non-cross resistant cytotoxic, has potential to offer a new regimen for the treatment of ovarian cancer in women who are refractory to standard drug regimens. Non-cross resistance to platinum is critical for the development of effective salvage regimens in this platinum resistant population. In addition bendamustine's cytotoxic effects are thought to occur via several mechanistic pathways, apoptosis, DNA repair, DNA replication, DNA transcription. The study seeks to determine the efficacy and safety of bendamustine in women with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary, fallopian tube cancer or primary peritoneal serous papillary carcinoma. Borderline ovarian tumors are not allowed.

2 Patients must have relapsed within 6 months of completing, or had a best response of increasing disease during any number of prior chemotherapy regimens with a platinum (either cisplatin or carboplatin) and a taxane (paclitaxel or docetaxel). These agents may have been administered concurrently or sequentially. Any number of additional regimens for recurrent disease will be allowed, as long as the patient performance status is 0-2 Gynecologic Oncology Group (GOG).

3 Patients must have measurable or evaluable (i.e. positive serum Cancer Antigen (CA) -125 marker) disease. Scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration. Scans or ultrasounds for non -measurable disease must have been performed within 28 days prior to registration.

4 Prior radiation is allowed as long as it encompassed no more than 25% of the bone marrow. Debulking surgery for relapsed disease is allowed as long as the patient has measurable or evaluable disease remaining after the surgery. Patient must have recovered from all side effects of surgery.

5 Patients must not have received chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to registration. Patients must not have had a major surgery within 14 days prior to registration.

6 Patients must have a GOG performance status of 0-2.

7 Patients must have adequate liver function as defined by a serum bilirubin ≤2.0 x the institutional upper limit of normal (IULN), serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) ≤2.5 x the institutional upper limit of normal obtained within 14 days prior to registration.

8 Patients must have an adequate renal function as defined by a serum creatinine ≤1.5x the institutional upper limit of normal obtained within 14 days prior to registration

9 Patients must not have Class 3 /4 cardiac problems as defined by the New York Heart Association Criteria (e.g., congestive heart failure, myocardial infarction within 2 months of study)

10 Patients must not be pregnant or nursing as bendamustine maybe harmful to the developing fetus and newborn. Women of reproductive potential must have a negative serum pregnancy test within 7 days prior to registration. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.

11 No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

12 Patients must have the following hematological criteria: Hemoglobin of ≥9gm/dL White blood cell count ≥ 2500 Platelets ≥ 100,000

13 Patients must be ≥ 18 years of age.

-

Exclusion Criteria:

1. No borderline ovarian tumors and mixed mesodermal soft tissue sarcomas
2. No psychological, familial, sociological, or geographical conditions that do not permit medical follow-up or compliance with the study protocol
3. Except for cancer-related abnormalities, patients should not have unstable or preexisting major medical conditions
4. No medical life-threatening complications of their malignancies
5. No known severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, active uncontrolled infection, or HIV)
6. Inadequately controlled hypertension (defined as systolic blood pressure ≥ 150 and/or diastolic blood pressure ≥100 mmHg on antihypertensive medications)
7. New York Heart Association (NYHA) Grade III or greater congestive heart failure
8. Evidence of 5 to ≤10% loss of weight from baseline (baseline defined as the screening weight taken approximately 14 days of Day 0) that is not related to ascites or paracentesis.
9. Evidence of uncontrollable nausea
10. Presence of central nervous system or brain metastases
11. Known hypersensitivity to any component of bendamustine HCL

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Setsuko K Chambers, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine: Bendamustine Hydrochloride (HCL) 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
Period: Overall Study
Arm/Group | Bendamustine
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Primary Site [Number; unit: participants]
  Ovarian | 9
  Peritoneal | 1
Median number of prior regimens [Median (Full Range); unit: Regimens] | 5 [3 to 10]
Eastern Cooperative Oncology Group performance status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is a scale 0-5. A score of 0 indicates fully active, able to carry on all pre-disease performance without restriction; 1 indicates restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; For more information on the ECOG performance scale refer to Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.
  Participants
    0 | 9
    1 | 1
Tumor Grade [Number; unit: Participants] — Criteria met for determination of Grade:
  Grade 1: the least malignant, with well-differentiated cells Grade 2: intermediate, with moderately differentiated cells Grade 3: the most malignant, with poorly differentiated cells
  Participants
    2 | 2
    3 | 8
Cell Type [Number; unit: Participants]
  Serous | 6
  Endometrioid | 3
  Clear Cell | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival in Patients With Platinum and Taxane Refractory Ovarian Cancer, Fallopian Tube Cancer and Primary Peritoneal Cancer With Bendamustine Treatment.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria or Cancer Antigen (CA)125 response using the modified Gynecologic Cancer Intergroup(GCIG) criteria
Time Frame: life of the study
Measure: Median (Full Range); unit: Days
Groups:
- Bendamustine Median Progression Free Surivial in Months: bendamustine HCL 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
Arm/Group | Bendamustine Median Progression Free Surivial in Months
Number analyzed (Participants) | 10
Days | 140 [23 to 316]

2. Secondary Outcome: Toxicities of Patients Treated With Bendamustine.
Description: Grade 4 Toxicity
Time Frame: Life of the study
Measure: Number; unit: Partcipants
Groups:
- Bendamustine Grade 4 Toxicity: bendamustine HCL 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
Arm/Group | Bendamustine Grade 4 Toxicity
Number analyzed (Participants) | 10
Partcipants | 0

3. Primary Outcome: Overall Survival in Patients With Platinum and Taxane Refractory Ovarian Cancer, Fallopian Tube Cancer and Primary Peritoneal Cancer With Bendamustine Treatment.
Time Frame: Life of study
Measure: Median (Full Range); unit: Days
Groups:
- Median Overall Survival in Days: bendamustine HCL 90 mg/m2 intravenously on days 1(± 1 day) and 2 (± 1 day) every 28 days. If no grade ≥3 hematologic adverse event appears the dose will be escalated to 120 mg/m2 on days 1(± 1 day) and 2 (± 1 day) every 28 days at cycle 2.
Arm/Group | Median Overall Survival in Days
Number analyzed (Participants) | 10
Days | 393 [234 to 925]

ADVERSE EVENTS:
Time Frame: Life of study
Arm/Group | Bendamustine
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=10)
Small Bowel Obstruction (Gastrointestinal disorders) | 2 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine (N=10)
Fatigue (General disorders) | 4
Fever (General disorders) | 3
Rigors (General disorders) | 2
Weight Loss (General disorders) | 1
Hypotension (Cardiac disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Other (Skin and subcutaneous tissue disorders) | 1
Anoxeria (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dehydration (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Distention (General disorders) | 1
Dysgeusia (General disorders) | 3
Nausea (General disorders) | 6
Oral Mucositis (General disorders) | 2
Vomiting (General disorders) | 5
Other GI (Gastrointestinal disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 6
Neutrophils (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 5
Platlets (Blood and lymphatic system disorders) | 5
Cellulitis (Infections and infestations) | 1
Creatinine (Metabolism and nutrition disorders) | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypoantremia (Metabolism and nutrition disorders) | 1
Muscle weakness/ Cramping (Musculoskeletal and connective tissue disorders) | 2
Dizziness (General disorders) | 2
Sensory Neuropathy (General disorders) | 2
Pain Abdominal, chest, back (General disorders) | 3
Headache (General disorders) | 1
COugh/Dyspnea (General disorders) | 2

LIMITATIONS AND CAVEATS:
The team was not able to collect fresh tumor tissue at the time of the study, so we could not examine patient tumors to determine their DNA repair capabilities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No